CLINICAL TRIAL: NCT01076426
Title: The Clinical Use of Probiotics in the Uremia Patients Under Chronic Peritoneal Dialysis
Brief Title: Probiotics Use in the Chronic Peritoneal Dialysis Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Pro-bio Biotech Co. Ltd. (Industry)
Responsible Party: An-Bang Wu, MD, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HR-98-083
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-02

CONDITIONS: Peritonitis; Malnutrition
Keywords: probiotic; peritoneal dialysis; peritonitis; nutrition status
MeSH Terms: conditions — Peritonitis; Malnutrition | interventions — Oligosaccharides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotics (Experimental): probiotics treatment
  Interventions: Drug: Pro-biotics
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Oligosaccharide

INTERVENTIONS:
Drug: Pro-biotics — Pro-biotics and placebo one pack per day is given to the two group. And then evaluate the peritonitis rate and nutrition status.
  Arms: Probiotics
Dietary Supplement: Oligosaccharide — oligosaccharide one pack per day
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether probiotics can improve the nutrition status and prevent peritonitis in the chronic peritoneal dialysis patients.

DETAILED DESCRIPTION:
Peritoneal dialysis was one of therapies for uremia patient. However, peritoneal dialysis related peritonitis was a major complication for these patients. Severe and prolong peritonitis may led to membrane failure and drop out of peritoneal dialysis. Among the pathogens, G(+) bacteria came from skin surface and G(-) bacteria came from gastrointestinal tract. The later might be related to the pathogens in the gastrointestinal tract, and led to peritonitis if constipation or diarrhea developed. In addition, intestinal pathogens may be related to chronic inflammation in uremia patients. There was a MIA syndrome (malnutrition, inflammation and atherosclerosis) noted before, and chronic inflammation may be related to malnutrition. Today, we know that nutrition status and inflammation marker (CRP) may be associated with patients' outcome. Many gastrointestinal syndromes such as constipation suffer our patients. The dialysate in the abdominal cavity may further exacerbate the appetite. The probiotics was though to improve the pathogens in intestinal tract, improve gastrointestinal function. We want to decrease the incidence of peritonitis by using the probiotics. In addition, the improvement in gastrointestinal function can increase the nutrition status.

ELIGIBILITY:
Inclusion Criteria:

* 1. uremia patient under chronic peritoneal dialysis ≧ 3 months
* 2. Age between 16 and 75 years

Exclusion Criteria:

* 1. uremia patient with advanced malignance disease
* 2. uremia patient had more than 2 episode of G(+) peritonitis within the last one year
* 3. uremia patient with expected life ≦ 1 years
* 4. uremia patient with the history of drug or alcohol abuse
* 5. uremia patient with poor drug compliance
* 6. uremia patient with active infection disease
* 7. uremia patient with uncontrolled autoimmune disease such as SLE

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
peritonitis rate | one year
nutrition status | 3, 6, 9, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: An-Bang WU, MD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan, Taiwan